CLINICAL TRIAL: NCT03085199
Title: Laparoscopic Reinforcement Suture (LARS) on Staple-line of Duodenal Stump Using Barbed Suture in Laparoscopic Gastrectomy for Gastric Cancer: A Prospective Single Arm Phase II Study
Brief Title: Laparoscopic Reinforcement Suture (LARS) of Duodenal Stump A Prospective Single Arm Phase II Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Kwan Woo Kim, Director, Dong-A University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAUHIRB-16-010
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Duodenal Stump Leak
Keywords: gastric cancer; laparoscopic gastrectomy; laparoscopic reinforcement suture (LARS)
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic reinforcement suture (Other): After cutting of duodenal stump of about 2 cm length using linear stapler, laparoscopic reinforcement suture commenced from upper to lower part on staple-line of duodenal stump. Continuous suture with invagination was performed using a barbed suture. In case of patient with short duodenal stump because of chronic ulcer or ectopic pancreas at duodenal bulb, 2 or 3 interrupted sutures without invagination of duodenal stump was conducted using barbed sutures.
  Interventions: Procedure: Laparoscopic reinforcement suture

INTERVENTIONS:
Procedure: Laparoscopic reinforcement suture — After cutting of duodenal stump of about 2 cm length using linear stapler, LARS commenced from upper to lower part on staple-line of duodenal stump. Continuous suture with invagination was performed using a barbed suture. In case of patient with short duodenal stump because of chronic ulcer or ectopic pancreas at duodenal bulb, 2 or 3 interrupted sutures without invagination of duodenal stump was conducted using barbed sutures.

SUMMARY:
Until now, no prospective clinical trial for duodenal stump leakage after laparoscopic or open gastrectomy for gastric cancer patients has been conducted.

We already introduced a technique of laparoscopic reinforcement suture (LARS) on staple-line of duodenal stump using barbed suture for prevention of duodenal stump leakage. Therefore, a prospective phase II study was designed for safety of this technique.

DETAILED DESCRIPTION:
As the results of recent prospective randomized controlled clinical trials, laparoscopic gastrectomy has been accepted by one of standard treatments for early gastric cancer in Korea, Japan and China.

However, duodenal stump leakage remains one of the fetal complications after gastrectomy until now. The incidence of duodenal stump leakage is reportedly between 1.6% to 5% in Billroth II or Roux en Y reconstruction after gastrectomy for gastric cancer. According to a recent multicenter study, the laparoscopic approach increased the risk of duodenal stump leakage development comparing to open approach.

Until now, no prospective clinical trial for duodenal stump leakage after laparoscopic or open gastrectomy for gastric cancer patients has been conducted. I already introduced a technique of laparoscopic reinforcement suture (LARS) on staple-line of duodenal stump using barbed suture for prevention of duodenal stump leakage. Therefore, a prospective phase II study was designed for safety of this technique.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven gastric adenocarcinoma that were treated with laparoscopic distal or total gastrectomy and B-II or Roux en Y reconstruction and age of above 19 years

Exclusion Criteria:

* history of previous abdominal surgery except cholecystectomy and would be performed combined abdominal surgery except cholecystectomy. And also patients with advanced gastric cancer with gastric outlet obstruction or cancer invasion to pylorus

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of duodenal stump fistula within postoperative 30 days | 30 days
  Duodenal stump fistula was defined as clinical suspicion, laboratory finding of fluid from drain or radiologic finding such as CT scan or fistulogram.

CONTACTS AND LOCATIONS:
Overall Officials: kwan woo kim, phd, Principal Investigator — Dong-A University Hospital
Locations (1):
- University of Inje College of Medicine, Haeundae Paik Hopsital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ali BI, Park CH, Song KY. Outcomes of Non-Operative Treatment for Duodenal Stump Leakage after Gastrectomy in Patients with Gastric Cancer. J Gastric Cancer. 2016 Mar;16(1):28-33. doi: 10.5230/jgc.2016.16.1.28. Epub 2016 Mar 31. PMID 27104024